CLINICAL TRIAL: NCT02237456
Title: Comparison of Intra Vascular Optical Coherence Tomography Systems for Assessment of Coronary Tissue, Metallic Stents and Bioresorbable Vascular Scaffolds - DOCTOR Compare
Brief Title: DOCTOR Compare - A Study in the "DOCTOR" Series (Does Optical Coherence Tomography Optimize Revascularization?"
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Niels Ramsing Holm, Doctor, Aarhus University Hospital Skejby
Other Study IDs: 1-10-72-59-14
Record Dates: First submitted 2014-06-24; First posted 2014-09-11 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Disease; Myocardial Infarction; Atherosclerosis
Keywords: Myocardial infarction; Atherosclerosis; PCI; OCT; Optical coherence tomography; Stent; Bioresorbable stents
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction; Atherosclerosis | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Comparison of OCT scans
Procedure: Comparison of Intra Vascular Optical Coherence Tomography Systems for Assessment of Coronary Tissue, Stents and Scaffolds - DOCTOR Compare

SUMMARY:
The purpose of this study is to compare optical coherence tomography (OCT) scans performed in the same coronary artery with two different OCT systems (Lunawave and OPTIS) before and after implantation of stents or bioresorbable scaffolds.

DETAILED DESCRIPTION:
Standard treatment of persons with narrowings of the heart's coronary artery is balloon treatment with implantation of stents (Percutaneous coronary intervention (PCI )). To evaluate disease in coronary arteries prior to, and during PCI , X-ray fluoroscopy with contrast is used. X-ray fluoroscopy produces little information of any disease changes in the vessel wall and implanted stents and especially polylactid acid (PLA) type bioresorbable scaffolds are visualized poorly .

Optical coherence tomography (OCT) is a light-based, high resolution, imaging modality for intra coronary assessment of tissue and implants. Currently two CE-marked OCT systems are used in clinical practice in (Illumien OPTIS, St. Jude Medical , Minnesota, USA and Lunawave, Terumo , Tokyo, Japan). It is a common assumption that the scanning images for the two systems are similar and are interpreted the same way.

The aim of the study is to assess if tissue, stents and PLA type scaffolds are presented with same characteristics by the two systems.

Same segment scans by the two systems will be systematically compared and reported.

Differences in scans by the two systems may have implications for the interpretation and thus may affect clinical decisions.

ELIGIBILITY:
Inclusion Criteria:

* Indication for intervention with PCI on the right or left coronary artery
* Age >18 years
* Must be able to give written informed consent

Exclusion Criteria:

* Expected life span of less than one year
* Pregnancy or possible pregnancy
* Cardiogenic shock
* Especially tortuous vessels
* Renal impairment (creatinine> 100 micromoles / L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing percutaneous coronary intervention (PCI) at Department of Cardiology, Aarhus University Hospital Skejby, will be invited to participate in the study. 12 patients will be included; 4 with acute ST-elevation myocardial infarct (STEMI) and 8 stable or stabilized patients.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Comparison of quantitative and semi-quantitative tissue analysis obtained with OCT images | Baseline
Characteristics of thrombic mass (average thickness of signal-rich area, shade degree) | Baseline
Characteristics of fibrous tissue (maximum scan penetrance) | Baseline
Characteristics of lipid plaque (signal intensities under the fibrous cap) | Baseline
Characteristics of calcium plaque (matched calcium plaques that can be quantified for sizes) | Baseline
Characteristics of vessel dissection (exploratory) | Baseline
Characteristics of the fibrous cap (minimum thickness) | Baseline

SECONDARY OUTCOMES:
Detection of stent struts | Baseline
  Stent evaluation obtained by Lunawawe recordings versus OPTIS recordings (including areas with thrombus, plaque, bare metal stent, bioresorbable stents, 3D reconstruction of stents (qualitative and quantitative assessment of stent visualization degree)

CONTACTS AND LOCATIONS:
Overall Officials: Niels R Holm, MD, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N, Denmark
  - Rigshospitalet, Copenhagen